CLINICAL TRIAL: NCT01041027
Title: A Pilot Phase II Trial of Radiation Therapy "Sandwiched" Between Paclitaxel and Carboplatin in Patients With High-Risk Endometrial Cancer After Standard Surgical Staging
Brief Title: Radiation Therapy, Paclitaxel, and Carboplatin in Treating Patients With High-Risk Endometrial Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to slow accrual. Results from the PORTEC3 the study rendered the hypothesis no longer valid.
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-03-060; NCI-2013-01224 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 07-062; NCI-2012-00458; 08-03-060 (Other: Albert Einstein College of Medicine); P30CA013330 (NIH)
Record Dates: First submitted 2009-12-29; First posted 2009-12-30 (Estimated); Results first posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Endometrial Adenocarcinoma; Stage IA Uterine Corpus Cancer; Stage IB Uterine Corpus Cancer; Stage II Uterine Corpus Cancer; Stage IIIA Uterine Corpus Cancer; Stage IIIB Uterine Corpus Cancer; Stage IIIC Uterine Corpus Cancer; Stage IVA Uterine Corpus Cancer; Stage IVB Uterine Corpus Cancer
MeSH Terms: interventions — Paclitaxel; Taxes; Carboplatin; Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (paclitaxel, carboplatin, radiation therapy) (Experimental): CHEMOTHERAPY (weeks 1-9, 13-21): Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for 3 courses during weeks 1-9 and 3 courses during weeks 13-21.
  RADIATION THERAPY (weeks 8-13 or 8-15): Patients with stage I disease undergo HDR brachytherapy once weekly for a total of 5 fractions during weeks 8-13. All other patients undergo EBRT QD 5 days a week for a total of 25 fractions during weeks 8-12 and HDR brachytherapy once weekly for a total of 3 fractions during weeks 13-15.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Radiation: Internal Radiation Therapy; Radiation: External Beam Radiation Therapy; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; TAX
Drug: Carboplatin — Given IV
Radiation: Internal Radiation Therapy — Undergo HDR brachytherapy
  Other Names: Brachytherapy; Internal Radiation; Internal Radiation Brachytherapy; Radiation Brachytherapy
Radiation: External Beam Radiation Therapy — Undergo EBRT
  Other Names: Definitive Radiation Therapy; EBRT; External Beam RT
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well radiation therapy, paclitaxel, and carboplatin work in treating patients with high-risk endometrial cancer. Radiation therapy uses high energy x rays to kill tumor cells. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing or by stopping them from spreading. Giving radiation therapy with chemotherapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate progression-free survival. II. To assess and document location of disease recurrence (distant vs local vs both) using this treatment regimen.

II. To evaluate the toxicity of radiation therapy "sandwiched" between cycles of paclitaxel/carboplatin chemotherapy in patients with high-risk endometrial cancer.

III. To evaluate the associations of cancer recurrence with tumor tissue expression levels of insulin-like growth factor-I (IGF-I), IGF-II, insulin-like growth factor binding protein 1 (IGFBP-1) and -3, insulin receptor, IGF-I receptor, estrogen receptor, and progesterone receptor.

OUTLINE:

CHEMOTHERAPY (weeks 1-9, 13-21): Patients receive paclitaxel intravenously (IV) over 3 hours and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for 3 courses during weeks 1-9 and 3 courses during weeks 13-21.

RADIATION THERAPY (weeks 8-13 or 8-15): Patients with stage I disease undergo high dose rate (HDR) brachytherapy once weekly for a total of 5 fractions during weeks 8-13. All other patients undergo external beam radiation therapy (EBRT) once daily (QD) 5 days a week for a total of 25 fractions during weeks 8-12 and HDR brachytherapy once weekly for a total of 3 fractions during weeks 13-15.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-documented high-risk endometrioid adenocarcinoma with no visible residual disease, defined by the following criteria:

  * Surgical stage I disease with < 50 myometrial invasion and grade 3 tumor (IAG3) with lymphovascular space involvement;
  * Surgical stage I disease with >= 50% myometrial invasion and grade 2 or 3 tumor (IBG2, IBG3);
  * Any surgical stage II disease (II);
  * Any surgical stage III disease (IIIA, IIIB, IIIC); and
  * Any surgical stage IV disease with no residual macroscopic tumor
* Surgical staging to include total abdominal hysterectomy, bilateral salpingo-oophorectomy, peritoneal washings, and lymph node samplings as per standard Gynecologic Oncology Group (GOG) criteria
* Eastern Cooperative Oncology Group (ECOG) performance status of < 2
* Written voluntary informed consent

Exclusion Criteria:

* Serum glutamic oxaloacetic transaminase (SGOT) and/or serum glutamate pyruvate transaminase (SGPT) > 2.5 times the institutional upper limit of normal
* Total serum bilirubin > 1.5 mg/dl
* History of chronic or active hepatitis
* Serum creatinine > 2.0 mg/dl
* Platelets < 100,000/mm^3
* Absolute neutrophil count (ANC) < 1500/mm^3
* Hemoglobin < 8.0 g/dl (the patient may be transfused prior to study entry)
* Patient has severe or uncontrolled concurrent medical disease (e.g. uncontrolled diabetes, unstable angina, myocardial infarction within 6 months, congestive heart failure, etc.)
* Patient with any prior chemotherapy or radiotherapy for pelvic malignancy
* Patients with dementia or altered mental status that would prohibit the giving and understanding of informed consent at the time of study entry
* Patients with any history of cancer with the exception of non-melanoma skin cancer are excluded if there is any evidence of other malignancy being present within the past five years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-01-16 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Yi-Shin Kuo, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 31 participants were enrolled into the study between 1/16/2009 (date the first participant was enrolled) and 6/3/2019 (date final participant was enrolled)
Pre-assignment Details: 40 participants were recruited. Of the 40 participants, 1 participant was not consented and 8 participants screen failed. 31 participants were enrolled and randomized into the study.
Groups:
- Treatment (Paclitaxel, Carboplatin, Radiation Therapy): CHEMOTHERAPY (weeks 1-9, 13-21): Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for 3 courses during weeks 1-9 and 3 courses during weeks 13-21.
  RADIATION THERAPY (weeks 8-13 or 8-15): Patients with stage I disease undergo HDR brachytherapy once weekly for a total of 5 fractions during weeks 8-13. All other patients undergo EBRT QD 5 days a week for a total of 25 fractions during weeks 8-12 and HDR brachytherapy once weekly for a total of 3 fractions during weeks 13-15.
  Paclitaxel: Given IV
  Carboplatin: Given IV
  Internal Radiation Therapy: Undergo HDR brachytherapy
  External Beam Radiation Therapy: Undergo EBRT
  Laboratory Biomarker Analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Paclitaxel, Carboplatin, Radiation Therapy)
Started | 31
Completed | 23
Not Completed | 8
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Violation | 1
Not completed — Delayed Radiation Therapy | 1
Not completed — Adverse Event | 4

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Paclitaxel, Carboplatin, Radiation Therapy)
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 12
  More than one race | 2
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS will be analyzed using standard survival analytic methods, including the Kaplan-Meier approach for estimating the survival distribution. Median time to progression and 95% confidence intervals will be estimated from the Kaplan-Meier curves.
Time Frame: From randomization until documented tumor recurrence or death from any cause, assessed up to 5 years
Population: PFS data was not collected and analyzed.
Arm/Group | Treatment (Paclitaxel, Carboplatin, Radiation Therapy)
Number analyzed (Participants) | 0

2. Secondary Outcome: Expression Levels of IGF-1
Description: Associations of PFS with tumor tissue expression levels of IGF-1 will be evaluated. Provided the number of events is sufficient, Cox proportional hazards models will be fit to the data to explore these associations.
Time Frame: Up to 5 years
Population: IGF-1 expression data was not collected and analyzed.
Arm/Group | Treatment (Paclitaxel, Carboplatin, Radiation Therapy)
Number analyzed (Participants) | 0

3. Secondary Outcome: Expression Levels of IGF-2
Description: Associations of PFS with tumor tissue expression levels of IGF-2 will be evaluated. Provided the number of events is sufficient, Cox proportional hazards models will be fit to the data to explore these associations.
Time Frame: Up to 5 years
Population: IGF-2 expression data was not collected and analyzed.
Arm/Group | Treatment (Paclitaxel, Carboplatin, Radiation Therapy)
Number analyzed (Participants) | 0

4. Secondary Outcome: Expression Levels of IGFBP-1
Description: Associations of PFS with tumor tissue expression levels of IGFBP-1 will be evaluated. Provided the number of events is sufficient, Cox proportional hazards models will be fit to the data to explore these associations.
Time Frame: Up to 5 years
Population: IGFBP-1 expression data was not collected and analyzed.
Arm/Group | Treatment (Paclitaxel, Carboplatin, Radiation Therapy)
Number analyzed (Participants) | 0

5. Secondary Outcome: Expression Levels of IGFBP-3
Description: Associations of PFS with tumor tissue expression levels of IGFBP-3 will be evaluated. Provided the number of events is sufficient, Cox proportional hazards models will be fit to the data to explore these associations.
Time Frame: Up to 5 years
Population: IGFBP-3 expression data was not collected and analyzed.
Arm/Group | Treatment (Paclitaxel, Carboplatin, Radiation Therapy)
Number analyzed (Participants) | 0

6. Secondary Outcome: Expression Levels of Insulin Receptor
Description: Associations of PFS with tumor tissue expression levels of insulin receptor will be evaluated. Provided the number of events is sufficient, Cox proportional hazards models will be fit to the data to explore these associations.
Time Frame: Up to 5 years
Population: Insulin receptor expression data was not collected and analyzed.
Arm/Group | Treatment (Paclitaxel, Carboplatin, Radiation Therapy)
Number analyzed (Participants) | 0

7. Secondary Outcome: Expression Levels of IGF-1 Receptor
Description: Associations of PFS with tumor tissue expression levels of IGF-1 receptor will be evaluated. Provided the number of events is sufficient, Cox proportional hazards models will be fit to the data to explore these associations.
Time Frame: Up to 5 years
Population: IGF-1 receptor expression data was not collected and analyzed.
Arm/Group | Treatment (Paclitaxel, Carboplatin, Radiation Therapy)
Number analyzed (Participants) | 0

8. Secondary Outcome: Expression Levels of Estrogen Receptor
Description: Associations of PFS with tumor tissue expression levels of estrogen receptor will be evaluated. Provided the number of events is sufficient, Cox proportional hazards models will be fit to the data to explore these associations.
Time Frame: Up to 5 years
Population: Estrogen receptor expression data was not collected and analyzed.
Arm/Group | Treatment (Paclitaxel, Carboplatin, Radiation Therapy)
Number analyzed (Participants) | 0

9. Secondary Outcome: Expression Levels of Progesterone Receptor
Description: Associations of PFS with tumor tissue expression levels of progesterone receptor will be evaluated. Provided the number of events is sufficient, Cox proportional hazards models will be fit to the data to explore these associations.
Time Frame: Up to 5 years
Population: Progesterone receptor expression data was not collected and analyzed.
Arm/Group | Treatment (Paclitaxel, Carboplatin, Radiation Therapy)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | Treatment (Paclitaxel, Carboplatin, Radiation Therapy)
All-Cause Mortality (participants affected / at risk) | 3/31
Serious Adverse Events (participants affected / at risk) | 2/31
Other Adverse Events (participants affected / at risk) | 5/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Paclitaxel, Carboplatin, Radiation Therapy) (N=31)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (4) — Grades 3-4
Anemia (Blood and lymphatic system disorders) | 2 (3)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) — Grade 4
Vaginal Hemorrhage (Reproductive system and breast disorders) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1) — Hospitalization for PICC site infection
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Paclitaxel, Carboplatin, Radiation Therapy) (N=31)
Anemia (Blood and lymphatic system disorders) | 4 (9)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (7)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2)
Alkaline Phosphatase Increased (Investigations) | 1 (2)
SGOT/SGPT ratio elevated (Investigations) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Increased ALT (Investigations) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Leukocytopenia (Blood and lymphatic system disorders) | 1 (2)
Leukopenia (Blood and lymphatic system disorders) | 1 (2)
Rash Acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Neuropathy (peripheral) (Nervous system disorders) | 3 (4)
Ankle Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Breast Pain (Reproductive system and breast disorders) | 1 (2)
Neutrophil Count Decreased (Investigations) | 1 (3)
Fatigue (General disorders) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Vulval Infection (Infections and infestations) | 1 (1)
Paresthesia (Nervous system disorders) | 2 (2) — Numbness
Mucositis (Gastrointestinal disorders) | 1 (1)
Pelvic Pain (Reproductive system and breast disorders) | 1 (1)
Finger Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Right hand
Proctitis (Gastrointestinal disorders) | 1 (2)
Vaginal Inflammation (Reproductive system and breast disorders) | 1 (1) — Inflammation lead to pain
Vaginal Irritation (Reproductive system and breast disorders) | 1 (1) — Verbatim term
Upper Respiratory Infection (Infections and infestations) | 1 (1)
Cystitis (Renal and urinary disorders) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (1)
Hypertension (Vascular disorders) | 1 (4)
Toothache (Gastrointestinal disorders) | 1 (1)
Skin Discoloration (Skin and subcutaneous tissue disorders) | 1 (1) — Verbatim term
Neutropenia (Blood and lymphatic system disorders) | 1 (1) — Verbatim term

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-22): https://cdn.clinicaltrials.gov/large-docs/27/NCT01041027/Prot_SAP_000.pdf